CLINICAL TRIAL: NCT05458011
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study With an Open-Label Treatment Period of Fremanezumab Administered Subcutaneously Monthly or Quarterly for the Preventive Treatment of Migraine in Adult Chinese Patients
Brief Title: A Randomized, Double-Blind, Placebo-Controlled Study With an Open-Label Period on Efficacy and Safety of Fremanezumab in Chinese Adults With Migraine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TV48125-CNS-30088
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab; erenumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fremanezumab Monthly (Experimental): Double Blind (DB) Period: Participants will receive fremanezumab once a month (approximately every 4 weeks). Participants will receive a single injection of fremanezumab and two placebo injections on Day 1, and a single injection of fremanezumab on Days 29 and 57.
  Open Label (OL) Period: Participants will receive fremanezumab once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Fremanezumab Quarterly (Experimental): DB Period: Participants will receive fremanezumab once a quarter (once at the beginning of the 12-week double-blind treatment period). Participants will receive 3 injections of fremanezumab on Day 1, and a single placebo injection on Days 29 and 57.
  OL Period: Participants will receive fremanezumab once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
  Interventions: Drug: Fremanezumab; Drug: Placebo
- Placebo (Placebo Comparator): DB Period: Participants will receive placebo once a month (approximately every 4 weeks). Participants will receive 3 placebo injections on Day 1, and a single injection of placebo on Days 29 and 57.
  OL Period: Participants will receive fremanezumab once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fremanezumab — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection
  Other Names: TEV-48125; Ajovy
  Arms: Fremanezumab Monthly; Fremanezumab Quarterly
Drug: Placebo — Pharmaceutical form: solution for injection
  Route of administration: subcutaneous injection

SUMMARY:
Primary Objective:

To demonstrate the efficacy of fremanezumab administered as monthly and quarterly subcutaneous (sc) injections to adult Chinese participants with migraine.

Secondary Objectives:

* To further demonstrate the efficacy of fremanezumab administered as monthly and quarterly sc injections.
* To evaluate the safety and tolerability of fremanezumab administered as monthly and quarterly sc injections.

DETAILED DESCRIPTION:
The total study duration for participants is planned to be approximately 9 months. The study will consist of a screening visit, a baseline period (4 weeks), a 12-week double-blind treatment period, a 12-week open-label treatment period, and a follow-up period lasting approximately 3 months after the last dose of treatment.

ELIGIBILITY:
Inclusion Criteria:

* The participant has a diagnosis of migraine with onset at ≤50 years of age.
* The participant has a body weight ≥45 kg and body mass index within the range 17.5 to 34.9 kg/m2 (inclusive).
* The participant has a history of migraine for ≥12 months prior to screening.
* Women of childbearing potential (WOCBP) whose male partners are potentially fertile (that is; no vasectomy) must use highly effective birth control methods for the duration of the study and for 6.0 months after discontinuation of investigational medicinal product (IMP).
* Men must be sterile or, if they are potentially fertile/reproductively competent (not congenitally sterile) and their female partners are of childbearing potential, should use highly effective birth control for the duration of the study.
* Additional criteria apply, please contact the investigator for more information.

Exclusion Criteria:

* Use of medications containing opioids (including codeine), barbiturates (including butalbital), or any combination product containing opioids or barbiturates (including butalbital) on more than 4 days during the screening period for the treatment of migraine or for any other reason.
* Has used an intervention/device (eg, scheduled nerve blocks or transcranial magnetic stimulation) for migraine, or in the head or neck area, during the 2 months prior to screening (visit 1).
* History of clinically significant cardiovascular disease or vascular ischemia (such as myocardial, neurological [eg, cerebral ischemia], or peripheral extremity ischemia or other ischemic event) or thromboembolic events (arterial or venous thrombotic or embolic events), such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism.
* History of human immunodeficiency virus, tuberculosis, Lyme disease, or a known or suspected active infection of coronavirus disease 2019 (COVID-19).
* Known current infection or history of infection in the past 6 months with hepatitis B or C viruses.
* History of cancer in the past 5 years, except for appropriately treated non-melanoma skin carcinoma.
* History of hypersensitivity reactions to injected proteins, including monoclonal antibodies (mAbs), or a history of Stevens-Johnson Syndrome or toxic epidermal necrolysis syndrome, or is concomitantly using lamotrigine.
* Any clinically significant uncontrolled medical condition (treated or untreated).
* History of alcohol or drug abuse during the past 2 years or drug dependence during the past 5 years.
* Additional criteria apply, please contact the investigator for more information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (29):
- China (29):
  - Teva Investigational Site 88028, Baotou Shi
  - Teva Investigational Site 88004, Beijing
  - Teva Investigational Site 88001, Beijing
  - Teva Investigational Site 88008, Changchun
  - Teva Investigational Site 88009, Changchun
  - Teva Investigational Site 88022, Changsha Shi
  - Teva Investigational Site 88030, Changsha Shi
  - Teva Investigational Site 88003, Chengdu
  - Teva Investigational Site 88029, Chongqing
  - Teva Investigational Site 88019, Fuzhou
  - Teva Investigational Site 88020, Guangzhou
  - Teva Investigational Site 88013, Guiyang
  - Teva Investigational Site 88026, Harbin
  - Teva Investigational Site 88010, Lianyungang
  - Teva Investigational Site 88005, Luoyang
  - Teva Investigational Site 88033, Rizhao
  - Teva Investigational Site 88021, Shanghaishi
  - Teva Investigational Site 88025, Shanghaishi
  - Teva Investigational Site 88016, Shenyang
  - Teva Investigational Site 88011, Shijiazhuang
  - Teva Investigational Site 88015, Suzhou
  - Teva Investigational Site 88024, Tianjin
  - Teva Investigational Site 88023, Tianjin
  - Teva Investigational Site 88017, Wenzhou
  - Teva Investigational Site 88012, Wuhan
  - Teva Investigational Site 88006, Wuhan
  - Teva Investigational Site 88032, Xining
  - Teva Investigational Site 88031, Zhanjiang
  - Teva Investigational Site 88034, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol and the statistical analysis plan. Requests will be reviewed for scientific merit, product approval status, and conflicts of interest. Patient level data will be de-identified and study documents will be redacted to protect the privacy of trial participants and to protect commercially confidential information. Please email USMedInfo@tevapharm.com to make your request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 454 participants were screened; of which 365 participants were randomized and included in the analysis.
Groups:
- Placebo: Double-blind (DB) Period: Participants received placebo subcutaneously (SC) once a month (approximately every 4 weeks). Participants received 3 placebo injections on Day 1, and a single injection of placebo on Days 29 and 57.
  Open-label (OL) Period: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
- Fremanezumab Monthly: DB Period: Participants received fremanezumab SC once a month (approximately every 4 weeks). Participants received a single injection of fremanezumab and two placebo injections on Day 1, and a single injection of fremanezumab on Days 29 and 57.
  OL Period: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
- Fremanezumab Quarterly: DB Period: Participants received fremanezumab SC once a quarter (once at the beginning of the 12-week DB treatment period). Participants received 3 injections of fremanezumab on Day 1, and a single placebo injection on Days 29 and 57.
  OL Period: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
Period: DB Period (12 Weeks)
Arm/Group | Placebo | Fremanezumab Monthly | Fremanezumab Quarterly
Started | 183 | 91 | 91
DB Safety Analysis Set (All randomized participants who received at least 1 dose of study drug during the DB treatment period.) | 183 | 91 | 91
DB Modified ITT (mITT) Analysis Set (All randomized participants who received at least 1 dose of study drug during the DB treatment period and had ≥10 days of postbaseline efficacy assessment on primary endpoint.) | 182 | 90 | 89
Completed | 177 | 87 | 86
Not Completed | 6 | 4 | 5
Not completed — Adverse Event | 2 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Non-compliance with trial drug | 0 | 0 | 1
Not completed — Protocol deviation | 0 | 2 | 2
Period: OL Period (12 Weeks)
Arm/Group | Placebo | Fremanezumab Monthly | Fremanezumab Quarterly
Started | 175 (2 participants who completed the DB treatment period did not rollover to the OL treatment period.) | 86 (1 participant who completed the DB treatment period did not rollover to the OL treatment period.) | 85 (1 participant who completed the DB treatment period did not rollover to the OL treatment period.)
OL Safety Analysis Set (All randomized participants who received at least 1 dose of study drug during the OL treatment period.) | 175 | 86 | 85
Completed | 174 | 81 | 84
Not Completed | 1 | 5 | 1
Not completed — Adverse Event | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) analysis set included all randomized participants.
Groups:
- Placebo: DB Period: Participants received placebo SC once a month (approximately every 4 weeks). Participants received 3 placebo injections on Day 1, and a single injection of placebo on Days 29 and 57.
  OL Period: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
- Total: Total of all reporting groups
Arm/Group | Placebo | Fremanezumab Monthly | Fremanezumab Quarterly | Total
Number analyzed (Participants) | 183 | 91 | 91 | 365
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (10.03) | 38.6 (9.42) | 39.7 (10.89) | 38.9 (10.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 71 | 73 | 286
  Male | 41 | 20 | 18 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 183 | 91 | 90 | 364
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 183 | 91 | 91 | 365
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of Migraine Days [Mean (Standard Deviation); unit: days] — A migraine day was defined as a calendar day where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for migraine with or without aura or; a calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine specific medications (triptans and ergot compounds).
  days | 11.0 (4.96) | 10.4 (5.94) | 10.4 (5.20) | 10.7 (5.27)

OUTCOME MEASURES:

1. Primary Outcome: Double Blind (DB) Period: Mean Change From Baseline in Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as a calendar day where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for migraine with or without aura or; a calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28. Least square (LS) mean was calculated using analysis of covariance (ANCOVA).
Time Frame: Baseline (Day -28 to Day -1), up to Week 12
Population: DB mITT analysis set included participants who received at least 1 dose of study drug and had at least 10 days of postbaseline efficacy assessment on the primary endpoint. Efficacy analysis was planned to be evaluated combined for both fremanezumab dose treatment groups.
Measure: Least Squares Mean (Standard Error); unit: days/month
Groups:
- Placebo: Participants received placebo SC once a month (approximately every 4 weeks). Participants received 3 placebo injections on Day 1, and a single injection of placebo on Days 29 and 57.
- Fremanezumab Monthly/Quarterly: Participants received fremanezumab SC once a month (approximately every 4 weeks) or once a quarter (once at the beginning of the 12-week DB treatment period).
  Participants received a single injection of fremanezumab and two placebo injections on Day 1, and a single injection of fremanezumab on Days 29 and 57 during Fremanezumab Monthly schedule.
  Participants received 3 injections of fremanezumab on Day 1, and a single placebo injection on Days 29 and 57 during Fremanezumab quarterly schedule.
Arm/Group | Placebo | Fremanezumab Monthly/Quarterly
Number analyzed (Participants) | 182 | 179
days/month | -2.8 (0.48) | -4.6 (0.48)
Statistical Analysis 1: Comparison: Placebo vs Fremanezumab Monthly/Quarterly; Test type: Other; p < 0.0001, ANCOVA; LS Mean Difference = -1.8, 95% CI 2-sided [-2.66 to -0.95], Standard Error of Mean 0.44

2. Secondary Outcome: DB Period: Mean Change From Baseline in the Average Number of Migraine Days During the 4-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as a calendar day where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for migraine with or without aura or; a calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 4-week period/number of days with assessments recorded in e-diary for 4-week period) * 28.
Time Frame: Baseline (Day -28 to Day -1), Up to Week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days
Arm/Group | Placebo | Fremanezumab Monthly/Quarterly
Number analyzed (Participants) | 182 | 179
days | -2.2 (0.52) | -4.5 (0.52)

3. Secondary Outcome: DB Period: Mean Change From Baseline in the Monthly Average Number of Days of Use of Any Acute Headache Medications During the 12-Week Period After the First Dose of Fremanezumab
Description: Participants recorded any headache medications (name of drug, number of tablets/capsules, and the dose in milligrams per tablet/capsule) taken each day in their electronic headache diary device. Acute headache medication included opioids, barbiturates, triptans, ergots, non-steroidal anti-inflammatory drugs (NSAIDs), acetaminophen and their combination products. Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28.
Time Frame: Baseline (Day -28 to Day -1), Up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Monthly/Quarterly
Number analyzed (Participants) | 182 | 179
days/month | -1.1 (0.41) | -3.0 (0.41)

4. Secondary Outcome: DB Period: Number of Participants Reaching at Least 50% Reduction From Baseline in Monthly Average Number of Migraine Days During the 12-Week Period After the First Dose of Fremanezumab
Description: A migraine day was defined as a calendar day where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for migraine with or without aura or; a calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of a headache meeting the criteria for probable migraine, a migraine subtype where only 1 migraine criterion is missing; a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine specific medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28.
Time Frame: Baseline (Day -28 to Day-1), Up to Week 12
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Monthly/Quarterly
Number analyzed (Participants) | 182 | 179
Participants | 63 | 103

5. Secondary Outcome: DB Period: Mean Change From Baseline in the Monthly Average Number of Headache Days of at Least Moderate Severity During the 12-Week Period After the First Dose of Fremanezumab
Description: A headache day of at least moderate severity was defined as a calendar day (00:00 to 23:59) where the participant reported either of the following: A calendar day (0:00 to 23:59) demonstrating at least 2 consecutive hours of headache of at least moderate severity; or a calendar day (0:00 to 23:59) demonstrating a headache of any duration that was treated with migraine-specific acute medications (triptans and ergot compounds). Monthly averages were derived and normalized to 28 days equivalent by formula: (number of days of efficacy variable over 12-week period/number of days with assessments recorded in e-diary for 12-week period) * 28.
Time Frame: Baseline (Day -28 to Day -1), Up to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: days/month
Arm/Group | Placebo | Fremanezumab Monthly/Quarterly
Number analyzed (Participants) | 182 | 179
days/month | -2.4 (0.43) | -4.5 (0.43)

6. Secondary Outcome: DB Period: Number of Participants With At Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious AEs (SAEs) were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that occurred after the first dose of study drug was administered through end of the trial. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 0 up to Week 12
Population: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- DB Period: Placebo: Participants received placebo SC once a month (approximately every 4 weeks). Participants received 3 placebo injections on Day 1, and a single injection of placebo on Days 29 and 57.
- DB Period: Fremanezumab Monthly: Participants received fremanezumab SC once a month (approximately every 4 weeks). Participants received a single injection of fremanezumab and two placebo injections on Day 1, and a single injection of fremanezumab on Days 29 and 57.
- DB Period: Fremanezumab Quarterly: Participants received fremanezumab SC once a quarter (once at the beginning of the 12-week DB treatment period). Participants received 3 injections of fremanezumab on Day 1, and a single placebo injection on Days 29 and 57.
Arm/Group | DB Period: Placebo | DB Period: Fremanezumab Monthly | DB Period: Fremanezumab Quarterly
Number analyzed (Participants) | 183 | 91 | 91
Participants | 79 | 48 | 37

7. Secondary Outcome: DB Period: Number of Participants Who Did Not Complete the Study Due to AEs
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. TEAEs were defined as AEs that occurred after the first dose of study drug was administered through end of the trial. A summary of other non-serious AEs and all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: Week 0 up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Fremanezumab Monthly | DB Period: Fremanezumab Quarterly
Number analyzed (Participants) | 183 | 91 | 91
Participants | 2 | 1 | 1

8. Secondary Outcome: OL Period: Number of Participants With at Least One TEAE
Description: as for outcome 7
Time Frame: Week 12 up to Week 24
Population: The OL safety analysis set included all participants who received at least 1 dose of study drug during the OL treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- OL Period: Placebo/Fremanezumab; OL Period: Fremanezumab Monthly; OL Period: Fremanezumab Quarterly: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
Arm/Group | OL Period: Placebo/Fremanezumab | OL Period: Fremanezumab Monthly | OL Period: Fremanezumab Quarterly
Number analyzed (Participants) | 175 | 86 | 85
Participants | 78 | 40 | 38

9. Secondary Outcome: OL Period: Number of Participants Who Did Not Complete the Study Due to AEs
Description: as for outcome 7
Time Frame: Week 12 up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | OL Period: Placebo/Fremanezumab | OL Period: Fremanezumab Monthly | OL Period: Fremanezumab Quarterly
Number analyzed (Participants) | 175 | 86 | 85
Participants | 1 | 1 | 1

10. Secondary Outcome: DB Period: Number of Participants Who Received Concomitant Medications for AEs
Description: Concomitant medications included all medications taken while the participant was treated with the study drug. Any concomitant medication received by the participant for AEs was recorded on the case report form (CRF). Concomitant medications included: butalbital for migraine/headache, ergots for migraine/headache, NSAIDs for migraine/headache, NSAIDs for other reason than migraine/headache, opioids for migraine/headache, opioids for reasons other reason than migraine/headache, preventive medication as specified in the protocol for migraine/headache, preventive medication as specified in the protocol for other reason than migraine/headache, triptans for migraine/headache.
Time Frame: Week 0 up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Fremanezumab Monthly | DB Period: Fremanezumab Quarterly
Number analyzed (Participants) | 183 | 91 | 91
Participants | 51 | 28 | 23

11. Secondary Outcome: OL Period: Number of Participants Who Received Concomitant Medications for AEs
Description: as for outcome 10
Time Frame: Week 12 up to Week 24
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | OL Period: Placebo/Fremanezumab | OL Period: Fremanezumab Monthly | OL Period: Fremanezumab Quarterly
Number analyzed (Participants) | 175 | 86 | 85
Participants | 46 | 26 | 30

12. Secondary Outcome: Number of Participants With Treatment Emergent Anti-Drug Antibodies (ADA)
Time Frame: Day 1 up to Day 225
Population: Participants who received fremanezumab were analyzed for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Monthly | Fremanezumab Quarterly
Number analyzed (Participants) | 183 | 91 | 91
Participants | 28 | 11 | 9

13. Secondary Outcome: Number of Participants With Treatment-Emergent Neutralizing Antibodies (NAbs)
Time Frame: Day 1 up to Day 225
Population: Participants who received fremanezumab were analyzed for ADA.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Fremanezumab Monthly | Fremanezumab Quarterly
Number analyzed (Participants) | 183 | 91 | 91
Participants | 27 | 11 | 9

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 225
Description: DB safety analysis set included all randomized participants who received at least 1 dose of study drug during the DB treatment period. OL safety analysis set included all participants who received at least 1 dose of study drug during the OL treatment period.
Groups:
- OL Period: Placebo; OL Period: Fremanezumab Monthly; OL Period: Fremanezumab Quarterly: Participants received fremanezumab SC once a month (approximately every 4 weeks) administered as a single injection on Days 85, 113, and 141.
Arm/Group | DB Period: Placebo | DB Period: Fremanezumab Monthly | DB Period: Fremanezumab Quarterly | OL Period: Placebo | OL Period: Fremanezumab Monthly | OL Period: Fremanezumab Quarterly
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/91 | 0/91 | 0/175 | 0/86 | 0/85
Serious Adverse Events (participants affected / at risk) | 1/183 | 2/91 | 0/91 | 0/175 | 2/86 | 2/85
Other Adverse Events (participants affected / at risk) | 30/183 | 23/91 | 15/91 | 33/175 | 23/86 | 16/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=183) | DB Period: Fremanezumab Monthly (N=91) | DB Period: Fremanezumab Quarterly (N=91) | OL Period: Placebo (N=175) | OL Period: Fremanezumab Monthly (N=86) | OL Period: Fremanezumab Quarterly (N=85)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Placebo (N=183) | DB Period: Fremanezumab Monthly (N=91) | DB Period: Fremanezumab Quarterly (N=91) | OL Period: Placebo (N=175) | OL Period: Fremanezumab Monthly (N=86) | OL Period: Fremanezumab Quarterly (N=85)
Injection site erythema (General disorders) | 4 (4) | 5 (8) | 4 (5) | 5 (6) | 6 (12) | 3 (5)
Injection site pruritus (General disorders) | 1 (1) | 6 (9) | 3 (4) | 5 (5) | 5 (12) | 3 (8)
Injection site swelling (General disorders) | 6 (7) | 5 (7) | 2 (2) | 7 (9) | 6 (8) | 4 (6)
COVID-19 (Infections and infestations) | 6 (6) | 5 (5) | 2 (2) | 4 (4) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 17 (18) | 9 (9) | 7 (8) | 18 (20) | 8 (9) | 8 (11)
Hyperlipidaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5) | 3 (3) | 9 (9) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2023-03-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT05458011/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT05458011/SAP_001.pdf